CLINICAL TRIAL: NCT05379868
Title: Posterior Column Spinal Osteotomies in the Treatment of Adolescent Idiopathic Scoliosis. A Randomized Clinical Trial
Brief Title: Posterior Column Spinal Osteotomies in the Treatment of Adolescent Idiopathic Scoliosis
Acronym: ASPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other); Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Ilkka Helenius, Professor, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUS/3525/2021
Record Dates: First submitted 2022-03-23; First posted 2022-05-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Who Masked: Participant
Masking Description: Participants will not be informed of chosen treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Posterior column osteotomy (Active Comparator): Apical 3-5 posterior column osteotomies in addition to standard treatment
  Interventions: Procedure: Posterior column osteotomy
- No osteotomies (Placebo Comparator): Standard treatment
  Interventions: Procedure: No osteotomies

INTERVENTIONS:
Procedure: Posterior column osteotomy — Apical full facet joint resection. Study intervention does not involve a device.
  Other Names: Smith-Petersen osteotomy
  Arms: Posterior column osteotomy
Procedure: No osteotomies — Standard treatment
  Arms: No osteotomies

SUMMARY:
Background: Posterior column osteotomies (PCO) are routinely used to facilitate curve correction in surgical treatment of adolescent idiopathic scoliosis (AIS). Data regarding routine use of PCO is controversial, with conflicting data for coronal and sagittal plane correction and clinical benefit. Use of PCO has not been studied in the surgical treatment of AIS in a prospective randomized clinical trial.

Study Design: A randomized, multicenter clinical trial on children and adolescents undergoing posterior spinal fusion for idiopathic scoliosis using pedicle screw instrumentation. Sixty consecutive adolescents will be randomized into PCO or no PCO group after surgical exposure of the spine in 1:1 ratio.

Aims and Hypothesis: To compare PCO vs. no PCO groups for the correction of coronal and sagittal plane curve in children undergoing posterior spinal fusion for AIS. The investigators hypothesize that the correction of coronal curve and hypokyphosis will be better in PCO group without increasing blood loss or complications.

Inclusion criteria: Adolescents (aged 10 to 21 years of age) undergoing corrective surgery for idiopathic scoliosis using pedicle screw technique.

Exclusion criteria: Coagulation disorder, smoking, unwilling to consent, vertebral column resection, need for anteroposterior surgery.

Main outcome parameters: Primary outcome is the radiographic correction (Coronal and sagittal plane). Secondary outcomes include health-related quality of life (Scoliosis Research Society 24 outcome questionnaire), postoperative pain, rib hump, operative time, blood loss, hospital stay, and complications.

Ethical aspects: Ethical committee approval will be obtained. An informed consent will be obtained from all children and their parents.

Time schedule and budget: This study has ethical committee approval.There will be no extra costs as all information gathered will be part of normal surgical treatment of AIS. A part-time research nurse has been hired to take care of data collection into the database.

DETAILED DESCRIPTION:
Background AIS is the most common indication for major surgery in adolescents. The current standard of care for idiopathic scoliosis with a curve magnitude of over 40-50˚ is posterior spinal fusion (PSF) with pedicle screw fixation. Pedicle screws are implanted using posterior subperiostal approach into pedicles and vertebral bodies and the screws are then connected with longitudinal rods to allow correction of scoliosis. Spinal fusion is obtained by local bone graft on decorticated posterior spinal elements. 70% correction of scoliosis is expected with standard PSF surgery for idiopathic scoliosis (1).

Posterior osteotomies are used to facilitate correction of scoliosis during PSF. Concept of PCO was originally introduced in 1945 for treatment of spinal deformities in patients with rheumatoid arthritis and ankylosing spondylitis (2). Indications for use of PCO have later broadened to surgical correction of Scheuermann´s kyphosis and idiopathic scoliosis (3). Currently, the most commonly used technique was described by Ponte (4). In Ponte osteotomy a wide resection of the thoracic facet joints, laminae, and ligamentum flavum is conducted to generate a 5-10 mm posterior gap that closes with segmental instrumentation (4). Originally these osteotomies were utilized to correct hyperkyphotic deformities allowing approximately a 10-degree correction per spinal level (5). In AIS increase of curve correction up to 7%, and 15% correction of rip hump has been described with PCO (6). Up to 15% critical neuromonitoring changes have been observed in patients undergoing PCO (7). Although there is enhanced correction of the curve in AIS, no differences have been observed in patient reported outcome measures (PROM) (8). PCO is currently used to facilitate correction of AIS with reported enhancement of coronal and axial parameters. There are not any Level 1 studies evaluating the feasibility of PCO in the surgical treatment of AIS.

Aims and hypothesis To compare postoperative scoliosis, kyphosis, rib hump, hemoglobin and hematocrit decrease, length of hospital stay and complications in patients having PCO or not having PCO during posterior spinal fusion for AIS. The investigators hypothesize that patients with PCO have better correction of scoliosis with similar blood loss and complications.

Methods Study design - A randomized, clinical trial according to CONSORT criteria (9).

Patients - 60 adolescents undergoing posterior spinal fusion with pedicle screw instrumentation for idiopathic scoliosis will be randomized after exposure of the spine for PCO. PCO will be conducted at three adjacent levels at the apex of the curve.

Inclusion criteria - Patients will be included in the study if they fulfill the following criteria: between 10 and 21 years of age; no contraindication for PCO; suitable for posterior scoliosis surgery using all pedicle screw technique for AIS (thoracic scoliosis, Lenke classification Types 1 to 4); normal blood coagulation; a normal whole spine MRI except for the spinal deformity (juvenile or AIS).

Exclusion criteria - Need for anteroposterior surgery; the need for three column vertebral resection; smoking; diabetes mellitus or abnormalities in blood coagulation.

Randomization - Randomization to intervention and control groups (1:1) will be carried out using the sealed envelope technique at the time of completion of spinal exposure.

Outcomes - The main outcome measure is scoliosis and kyphosis correction and pulmonary function. Secondary outcome measures include rib hump correction, hemoglobin and hematocrit, blood loss (mls), drain output over 24 hours (mls), total blood loss (intra-operative blood loss + drain output); postoperative pain (NRS) and opioid consumption (48 hour oxycodone consumption), health related quality of life by SRS-24, and complications (intraoperative neuromonitoring change, neurologic deficit, cerebrospinal fluid leak).

Surgery - Surgical planning of implant placement and the need for the Ponte procedure will be carried out preoperatively. In case the correction is estimated to be insufficient without Ponte osteotomy, patient can be drawn from the study and Ponte osteotomy conducted according surgeon's judgement. Each patient will be placed in the prone position and the posterior elements will be exposed using electrocautery. Ponte osteotomy will be conducted as described previously (5). Briefly, after full facetectomies ligamentum flavum and laminae are resected for 5 mm are posteriorly at three adjacent levels. The deformity will be corrected using bilateral segmental pedicle screw instrumentation and en bloc vertebral column derotation. Spinal fusion is carried out using autograft acquired from facetectomies and osteotomies with bone graft extenders (iFactor, Cerapedics, Ic., Westminster, CO). Spinal cord monitoring (MEP, SSEP, lumbar nerve root EMG with or without pedicle screw stimulation) will be undertaken in all patients. A single subfascial drain (Hemovac Ch14; Zimmer, Warsaw, Indiana) will be placed and will be removed at 24 hours post-operatively. A sterile wound dressing will be applied at the end of surgery. All patients will be mobilized using a standardized protocol: sitting on the day of surgery, minimum four steps on 1st postoperative day, and progressively increasing walking distance with an aim to discharge patients on 4th -5 th postoperative day. Discharge criteria include ability to walk independently, no need for opioid prescription, and ability to empty bladder spontaneously without a significant urinary retention (>200 mL).

Anesthesia - All patients will have total intravenous anesthesia including dexmedetomidine, propofol and remifentanil-infusions. Mean arterial pressure between 65 mmHg and 75 mmHg during surgery and for the first 24 hours post-operatively. Cefuroxime will be used as antibiotic prophylaxis. All patients will receive PCA for 48 hours postoperatively along with long-acting Targiniq twice daily.

All patients will receive an intravenous bolus of tranexamic acid (30 mg/kg, maximum dose 1500 mg) within 30 minutes before incision and then an infusion (10 mg/kg/h, maximum dose 500 mg/h) during surgery. Intra-operative blood loss will be measured and recorded as the amount of blood collected in the cell saver, surgical wound dressings will be weighed during surgery, excluding any irrigation with saline. Allogenic red blood cells will be transfused if the Hb concentration goes below 80 g/L during surgery or during the hospital stay. Fresh frozen plasma will be given if the blood loss exceeds 50% of the patient's total blood volume. Platelets will be infused if the blood loss is more than 100% of the blood volume. The estimated blood volume will be calculated using a formula of 70 ml/kg x weight (kg) (12).

Statistical power - The sample-size requirement of 30 patients per group was calculated using a study power of 80%, a type I error (alpha) of 0.05, and an estimated effect size of 0.7. Effect size evaluation was based on the assumption that mean (SD) postoperative correction of scoliosis is 10 (14) degrees better in PCO group.

Ethical aspects Ethical committee approval will be obtained at our university hospital. All patients and their caregiver will provide a written informed consent to participate. Based on the surgeon's decision, a discontinuation of PCO surgery can be made, if there is any suspicion of complication due to PCO. The patient will remain in the intervention group for statistical comparison according to the intention-to-treat principle.

Time schedule This study will be started after ethical committee approval estimated in the beginning of 2022 and patient recruitment is estimated to be done by the end of 2025.

Budget Surgical treatment of adolescents with idiopathic scoliosis is according to the standard practice. There will be no extra costs due to this study. A part-time research nurse and PhD students will be hired using Valtion tutkimusrahoitus and external funding.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent idiopathic scoliosis (Lenke 1 to 4)
* Age at surgery between 10 and 21 years
* Cobb angle of 45 degrees or more
* Posterior spinal fusion

Exclusion Criteria:

* Anteroposterior surgery
* Vertebral column resection
* Smoking
* Diabetes mellitus
* Bleeding disorder

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Scoliosis correction | 2 year follow-up
  Cobb angle
Forced vital capacity | 2 year follow-up
  Lung volume
Kyphosis correction | 2 year follow-up
  Cobb angle

SECONDARY OUTCOMES:
Opioid consumption | 48 hours
  Pain outcome
SRS-24 total score | 2 year follow-up
  Health-Related Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Helenius, MD, PhD, Study Director — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No
Original data will be available only upon a reasonable request from the Principal Investigator at the time of publication

REFERENCES:
- [Background] Hresko MT. Clinical practice. Idiopathic scoliosis in adolescents. N Engl J Med. 2013 Feb 28;368(9):834-41. doi: 10.1056/NEJMcp1209063. No abstract available. PMID 23445094